CLINICAL TRIAL: NCT06852911
Title: The Diagnostic Significance of Exhaled Nitric Oxide (FeNO) With a Novel Technology in the Assessment of Bronchial Asthma
Brief Title: FeNO Detection in Asthma Diagnosis: A New Technology Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novlead Inc. (Industry)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: FeNO2403-1.3
Record Dates: First submitted 2025-02-14; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Bronchial Asthma; Airway Disease
Keywords: FeNO; Bronchial asthma; Tidal breathing
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asthma Patients (Other): 1. Individuals aged 18 years or older, regardless of gender;
  2. Patients who have been diagnosed with bronchial asthma in accordance with the international GINA 2023 diagnostic criteria;
  3. The presence of respiratory symptoms for a duration of no less than 6 weeks;
  4. A history of non-smoking or cessation of smoking for a period exceeding 5 years.
  Interventions: Diagnostic Test: Chemiluminescent FeNO Analyzer; Diagnostic Test: Electrochemical FeNO Analyzer
- Healthy (Other): 1. Participants must be at least 18 years of age, regardless of gender;
  2. There should be no documented history of allergic conditions or chronic respiratory illnesses, and no significant abnormalities should have been observed during physical examinations conducted in the preceding year;
  3. Individuals must not have experienced any acute illnesses, should not have a history of medication use, and must not exhibit typical symptoms of respiratory infections within the last four weeks;
  4. Participants must either have no history of smoking or must have ceased smoking for a duration exceeding five years.
  Interventions: Diagnostic Test: Chemiluminescent FeNO Analyzer; Diagnostic Test: Electrochemical FeNO Analyzer

INTERVENTIONS:
Diagnostic Test: Chemiluminescent FeNO Analyzer — A novel chemiluminescence FeNO Analyzer has been developed, capable of measuring both FeNO50 and FeNO during tidal breathing. Each participant underwent three testing sessions, with the results averaged, and the sequence of tests was randomized.
  Other Names: eNOglow
Diagnostic Test: Electrochemical FeNO Analyzer — Electrochemical FeNO analyzers are employed in clinical settings for the measurement of FeNO50. Each participant underwent three testing sessions, with the results averaged, and the sequence of tests was randomized.

SUMMARY:
The detection of exhaled nitric oxide (FeNO) represents a non-invasive, safe, and rapid approach for assessing endogenous nitric oxide (NO) levels within the airway. FeNO concentrations are closely associated with airway inflammation and hyperresponsiveness, and are currently recognized as biomarkers indicative of type II airway inflammation. Recent advancements in nitric oxide detection technology for both upper and lower airways, as well as for small and large airways, have provided significant insights for the diagnosis and management of conditions such as bronchial asthma, chronic cough, upper airway diseases, chronic obstructive pulmonary disease, and even rare airway disorders. Presently, FeNO measurement is frequently employed in the differential diagnosis and monitoring of airway inflammatory diseases.

The FeNO test is conducted using a FeNO test analyzer. Internationally, FeNO detection analyzers utilize three primary methodologies: chemiluminescence, laser, and electrochemical techniques. Among these, chemiluminescence is regarded as the "gold standard" globally. However, due to technical constraints, this methodology has not been clinically accessible within domestic settings. In China, the electrochemical FeNO analyzer is predominantly utilized, characterized by its compact size and portability. Nonetheless, this method necessitates patient cooperation during inhalation and exhalation, rendering it impractical for individuals who are unable to comply, such as children, the elderly, and severely ill patients. Consequently, FeNO detection poses significant challenges for these populations in China, representing a notable clinical gap.

The newly implemented technology employs an innovative domestic chemiluminescence FeNO analyzer, which is exclusively available in China. This analyzer, owing to its methodological advantages, is capable of obtaining FeNO detection values from patients' natural breathing patterns, facilitating rapid response and comprehensive FeNO assessment without requiring patient cooperation. This approach, referred to as the "Tidal-breathing of FeNO" enables the completion of FeNO assessments in patients who are unable to engage in inspiratory and expiratory maneuvers. This advancement is anticipated to enhance the diagnostic accuracy of airway inflammation in this demographic, thereby facilitating early diagnosis, precise treatment, and improved management of disease progression.

DETAILED DESCRIPTION:
1. Asthmatic patients and healthy individuals who fulfilled the inclusion criteria were categorized and assigned identification numbers.
2. The basic demographic and health-related information of the subjects was documented, including age, sex, height, weight, respiratory symptoms, medical history, allergy history, disease diagnosis, comorbidities, medication history, smoking history, lung function test results, and other relevant examinations.
3. Pre-testing requirements and preparations included:

   * Abstaining from all medications (including glucocorticoids, type II inflammatory monoclonal antibodies, leukotriene receptor antagonists, antihistamines, decongestants, hypertonic saline, bronchoconstrictor/diastolic agents, NO synthase inhibitors, and NO donor drugs such as nitroglycerin or L-arginine) for a duration of six hours prior to the test;

     * Fasting for three hours before the test;

       * Avoiding all forms of liquid intake (including alcohol and coffee), smoking (both active and passive), strenuous physical activity (such as running or aerobic exercise), and any respiratory diagnostic or therapeutic procedures (including pulmonary function tests and aerosol inhalation) for one hour prior to the test.
4. The researcher verified the subjects' compliance with the aforementioned testing requirements and proceeded with testing for those who met the criteria. Testing was uniformly scheduled during daytime hours.
5. Each participant underwent testing using both the moisture method and the online method, with the order of tests determined randomly via a randomization table to mitigate potential sequential effects. Each test was conducted in accordance with the ATS/ERS Technical Standard for the Determination of Exhaled Nitric Oxide (2005) and the operational guidelines for the equipment. Subjects were instructed to maintain an upright position and to repeat each test three times while in a resting state. A resting period of at least 30 seconds was mandated between tests, provided the subjects experienced no discomfort. The total duration of the testing procedure was anticipated to be approximately 20 minutes per individual.

ELIGIBILITY:
Patients:

Inclusion Criteria:

1. Participants must be a minimum of 18 years of age, irrespective of gender;
2. Individuals must possess a diagnosis of bronchial asthma that aligns with the international GINA 2023 diagnostic criteria;
3. Respiratory symptoms must have been evident for at least 6 weeks;
4. Participants should either have no history of smoking or have discontinued smoking for a period exceeding 5 years.

Exclusion Criteria:

1. The concurrent use of additional asthma medications (such as glucocorticoids) alongside short-acting bronchodilators within the prior 4 weeks;
2. A diagnosis of respiratory infection within the preceding 4 weeks;
3. Conditions such as pregnancy, lactation, or menstruation;
4. Participation in other clinical research studies;
5. Any underlying medical or psychiatric conditions that, in the investigator's assessment, would render the individual unsuitable for participation in the study.

Healthy:

Inclusion Criteria:

1. Participants must be at least 18 years of age, with no restrictions on gender;
2. Individuals should not have a history of allergic diseases or chronic respiratory conditions, and must not exhibit any significant abnormalities in health assessments conducted within the past year;
3. There should be no acute illnesses or medication history within the preceding four weeks, and participants must not display any typical symptoms of respiratory infections;
4. A history of smoking is not permitted, or individuals must have ceased smoking for a minimum of five years.

Exclusion Criteria:

1. Individuals who are pregnant, breastfeeding, or currently experiencing menstruation;
2. Those who have been on long-term medication;
3. Participants involved in other clinical research studies;
4. Any potential medical or psychological conditions that the researcher deems may render the subject unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Performance Assessment of FeNO Chemiluminescence Analyzer | Through study completion, an average of 6 months
  Assessment of the performance of the FeNO chemiluminescence analyzer, focusing on repeatability (coefficient of variation, CV), sensitivity, specificity, and receiver operating characteristic (ROC) curves

SECONDARY OUTCOMES:
Consistency Evaluation Between FeNO Analyzers | through study completion, an average of 6 months
  Evaluation of the consistency between the chemiluminescence FeNO analyzer and the electrochemical FeNO analyzers, utilizing correlation and Bland-Altman analysis.

OTHER OUTCOMES:
Cut-off of Tidal Breathing of FeNO | through study completion, an average of 6 months
  Analysis of the Tidal Breathing of FeNO for the chemiluminescence FeNO analyzer, employing the ROC method to identify the optimal cut-off value

CONTACTS AND LOCATIONS:
Overall Officials: Ailing Song, Principal Investigator — Wuxi Branch of Ruijin Hospital (Xinrui Hospital of Xinwu Distric, Wuxi)
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Wuxi Xinwu District Xinrui Hospital, Wuxi